CLINICAL TRIAL: NCT03868657
Title: The Physiological Effects of hERG Blockade on Metabolism
Brief Title: The Physiological Effects of Human Ether-a-go-go-Related Gene (hERG)Blockade on Metabolism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Signe Torekov (Other)
Responsible Party: Sponsor-Investigator, Signe Torekov, Associate Professor, University of Copenhagen
Organization: University of Copenhagen (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: H-1701307
Record Dates: First submitted 2019-01-27; First posted 2019-03-11 (Actual); Last update posted 2022-04-14 (Actual); Status verified 2022-04

CONDITIONS: Long QT Syndrome; Hypoglycemia
MeSH Terms: conditions — Long QT Syndrome; Hypoglycemia | interventions — Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Moxifloxacin (Active Comparator): Per os, 800 mg, once daily for 4 days
  Interventions: Drug: Moxifloxacin
- Placebo (Placebo Comparator): Per os, 800 mg, once daily for 4 days
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Moxifloxacin — Moxifloxacin is solely used to cause a known and for the drug well documented effect, namely blockade of the Kv11.1 channel.
  Arms: Moxifloxacin
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The human ether-a-go-go-related gene HERG (encoding Kv11.1 potassium channels) is expressed in different parts of the body including the heart, pancreas and intestines. In the heart, Kv11.1 channels play a role in ending depolarization by causing repolarization. Loss-of-function mutations of HERG cause long QT syndrome, a condition of elongated QT interval that can lead to ventricular tachycardia, syncope and sudden death. Kv11.1 channels are also found in pancreatic α- and β-cells and intestinal L-cells, where they seem to play a role in the secretion of insulin, glucagon and Glucagon-Like Peptide-1 (GLP-1). Carriers of loss-of-function mutations in the HERG gene have showed increased insulin and incretin responses after glucose ingestion and decreased fasting levels of glucagon compared to matched control persons. Blockade of Kv11.1 has shown to augment glucose dependent insulin secretion and decrease low-glucose stimulated glucagon secretion in isolated α- and β- cells. The investigators of this study hypothesize that a blockade of Kv11.1 channels will increase incretin and β cell function and decrease α cell function and thus lead to lower glucose levels in humans after glucose intake. To investigate this, The investigators of this study will perform a randomized, cross sectional study of up to 40 healthy study participants who will serve as their own controls. The study participants will undergo two 6-hours oral glucose tolerance tests, one after intake of a known Kv11.1 blocker (moxifloxacin) and one control oral glucose tolerance test after intake of placebo. Prior to both tests the study participants will wear a continuous glucose monitor and on the day of the tests they will fill out a glucose questionnaire. Investigation of the physiological role of HERG in metabolism may provide a better insight on metabolic regulation.

DETAILED DESCRIPTION:
Background and significance:

The human ether-a-go-go-related gene (HERG) encodes Kv11.1 voltage-gated potassium channels throughout different parts of the human body including the heart, pancreas and intestine. Potassium channels are important for ending the depolarization by causing repolarization in cells.

Hence, various mutations in HERG have effects on cardiac and metabolic functions. One known example in the case of loss-of-function mutations in HERG is a reduced outward flow of potassium during repolarization of the heart, leading to an elongated QT interval that can lead to ventricular tachycardia, cardiac syncope and sudden death - known as the long-QT syndrome (LQTS) (1, 2). LQTS caused by HERG mutations is the second most common type of LQTS (1).

With regards to metabolism, blockade of Kv11.1 has shown to augment glucose dependent insulin secretion (3-5) and decrease low-glucose stimulated glucagon secretion (4) in isolated β and α cells and to augment insulin secretion and reduce blood glucose in living mice(3).

A study of 11 patients with LQTS caused by HERG mutations showed that during a 6-hour OGTT, the mutation carriers experienced increased levels of insulin, GLP-1 and Gastric Inhibitory Polypeptide (GIP), decreased levels of glucose and lower fasting levels of glucagon compared to matched control persons(6).

In this study the investigators wish to investigate the effects of Kv11.1 blockade on incretin and insulin secretion and blood glucose levels after oral glucose intake in humans.

Research question Study hypothesis The investigators of this study hypothesize that Kv11.1 blockade will increase the metabolic response of serum insulin and GLP-1 (AUC/30 min) to a 6-hour 75 g oral glucose tolerance test (OGTT) in healthy individuals.

Objective To investigate the hypothesis, the investigators of this study want to examine the metabolic responses of up to 40 healthy test subjects to a 6-hours 75 g OGTT. The test subjects will serve as their own controls in a double-blinded crossover trial where they will undergo two 6-hours OGTTs separated by a 3 weeks washout period. During one OGTT they will have received moxifloxacin (800 mg/day), which is a known blocker of the Kv11.1 channel, and during the other OGTT they will have received placebo. Prior to and after the test the subjects will wear a continuous glucose monitor (CGM) and at the day of the test they will fill out a glucose questionnaire.

Moxifloxacin is solely used to cause a known and for the drug well documented effect, namely blockade of the Kv11.1 channel.

Study design:

A randomized controlled double-blinded crossover trial with up to 40 healthy participants, who will serve as their own controls. Study design is outlined in figure 1.

Screening visit (V0): At the screening visit, participants will:

* Be screened to assess their eligibility (anamnesis, weight/height measurements and 12-lead electrocardiography (ECG)). If found eligible:
* Be instructed to have a CGM monitor placed 4 days prior to test visit 1 (V1) for up to 7 days.
* Be randomized to either group A or B by a qualified unblinded person from the Department of Biomedical Sciences, University of Copenhagen:

  * Group A will first receive the active drug known to have Kv11.1 blockade effects (Moxifloxacin, 800 mg/day) 3 days prior to test visit 1 and then - after a 3 weeks wash-out period - receive a placebo drug prior to test visit 2.
  * Group B will first receive the placebo drug 3 days prior to test visit 1 and then - after a 3 weeks wash-out period - receive the active drug prior to test visit 2. Receive the drug for test visit 1 (Kv11.1 blocker or placebo) and be instructed to orally administer the drug every morning at 6.00 AM 3 days prior to and at the same morning as the test visit (V1). The unblinded person will make sure to provide the right drug to the participants.

Test visit 1 (V1): Participants will meet fasting since 10.00 PM the previous evening at 8.00 AM at the Department for Biomedical Sciences, University of Copenhagen.

* The participants will hand in a urine and fecal sample.
* A 75 g 6-hours oral glucose tolerance test (OGTT) will be performed. Crushed paracetamol, 1 g is added to the glucose mixture. Blood samples and ECGs will be drawn and collected together. Blood samples of 8 ml will be drawn at -20, -10, -0 minutes before and at 8, 15, 30, 45, 60, 75, 90, 105, 120, 135, 150, 180, 210, 240, 270, 300, 330, and 360 minutes after the glucose intake. All blood samples will be analyzed for hormones, glucose, electrolytes, plasma paracetamol, proteomics and metabolomics and from the -20 minutes sample DNA material will be extracted and used for genome analysis (not an extensive genome sequencing). The samples will be tested for mutations in genes associated with glucose metabolism in relation to obesity, diabetes and cardiovascular disease. HbA1c and lipids will be measured.
* Glucose questionnaires. Wash-out period: There will be a wash-out period of 3 weeks.
* Participants will come in and have a CGM monitor placed 4 days prior to test visit 2 (V2) for up to 7 days
* Participants will receive the drug (Kv11.1 blocker or placebo) and start to orally administer the drug every morning at the same time3 days prior to and at the same morning as the test visit 2.

Test visit 2 (V2): Same examinations as described for Visit 1.

Criteria for when tests can be performed:

* Participants have to have orally administered the study medication 3 days prior to and at the same morning as the test visits at the same time.
* Participants have to be fasting from 10hours before test visits. This includes foods, liquids, smoking, alcohol and medication (except Kv11.1 blocker and a small amount of water used for administration hereof)
* Participants are not allowed to perform any exercise the day before as well as the same morning as the test visit.
* Participant are not allowed to take paracetamol 24 hours before test visits. Unblinding: The randomization list will be stored on site at the Department of Biomedical Sciences at the University of Copenhagen. Subject number of the trial participant is matched with the list, which reveals to what group the participant is randomized. The unblinded person will perform any unblinding of the trial participants after Last Patient Last Visit.

Data Data management: The subject and the biological material obtained from the subject will be identified by subject number and trial identification number. Appropriate measures such as encryption or deletion will be enforced to protect the identity of human subjects in all presentations and publications as required by national requirements. Laboratory data will be transferred electronically from the laboratory performing clinical analyses and will be archived in secured hard drives with backup options. The electronic data will be considered source data. In cases where laboratory data is transferred via non-secure electronic networks, data will be encrypted during transfer. Data is saved for 20 years.

Source data: Source documents will be kept at the Department of Biomedical Sciences, University of Copenhagen. Source data registered directly in the Case Report Form (CRF) include anamnesis, weight and height measurements, ECG.

Evaluability for subjects for analysis: Withdrawn subjects will be replaced. Rescreening is allowed within the recruitment period, at the Investigator's discretion.

Statistical considerations Data analysis plan: To investigate whether Kv11.1 blockade significantly effects fasting and glucose-stimulated values of serum insulin and plasma glucagon, GLP-1, potassium and GIP concentrations, an ANOVA will be performed using age and sex as covariate, randomization group as independent variable and AUC change in serum insulin and plasma glucagon, GLP-1, potassium and GIP concentrations as dependent variables to examine if mean differences exist on study participants after intake of Kv11.1 blocker and without Kv11.1 blocker.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men and women
* Age ≥20 and ≤40 years
* BMI ≥18,5 and ≤27,5

Exclusion Criteria:

* Chronic diseases (cardiac, metabolic, liver) including a family history of congenital Long QT syndrome.
* QTc values >440 ms (men) and >450 ms (women)
* Clinical important and/or symptomatic bradycardia
* Regular medication (contraceptive pills allowed)
* Pregnancy and breastfeeding

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 44 (Actual)
Dates: Start 2019-01-28 (Actual); Primary Completion 2019-08-19 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Insulin and GLP-1 | First and second test day
  Change in serum insulin response (AUC/30 min) and GLP-1(AUC/30 min) to a 75 g oral glucose tolerance test between OGTT with and without Kv11.1 blocker (moxifloxacin).

SECONDARY OUTCOMES:
Glucose, Glucagon and GIP | First and second test day
  Change in plasma glucose, glucagon and GIP response to a 75g oral glucose tolerance test between OGTT with and without Kv11.1 blocker (moxifloxacin).
Continuous Glucose Monitor | First and second test day
  Change in CGM between OGTT with and without Kv11.1 blocker (moxifloxacin).

OTHER OUTCOMES:
Hypoglycemia questionnaires | First and second test day
  Change in hypoglycemia questionnaire frequency and severity score, where higher score are more frequent and severe, between OGTT with and without Kv11.1 blocker (moxifloxacin).
Electrolytes | First and second test day
  Change in plasma electrolytes levels between comparison of metabolomics patterns of the same individual
Gut microbiota | Baseline, after first test day, after second test day and after 6 months
  Changes in gut microbiota composition obtained from fecal samples
Acetaminophen | First and second test day
  Changes in serum acetaminophen AUC to a 75 g oral glucose tolerance test between OGTT with and without Kv11.1 blocker (moxifloxacin).

CONTACTS AND LOCATIONS:
Overall Officials: Signe S. Torekov, MSc, PhD, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Department of Biomedical Sciences, Copenhagen, Denmark